CLINICAL TRIAL: NCT03828370
Title: Smartphone Help for DWI Offenders and Their Families: A B-SMART App
Brief Title: DWI Offenders and Their Families App for Smartphones
Acronym: B-SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: University of New Mexico (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 0320; 2R44AA022850-02 (NIH)
Record Dates: First submitted 2019-01-31; First posted 2019-02-04 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Coping Skills; Family Relations

STUDY DESIGN:
Intervention Model Description: The B-SMART mobile web app will be evaluated in a randomized pretest-posttest controlled design. First-time DWI offenders and their CFMs will be randomized together to the intervention (B-SMART) or a usual and customary (UC) IID information condition comparison group (n=150) following baseline assessment.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual & Customary Information Group (Active Comparator): Study Cohort Assessment:
  Baseline 3 month follow-up/ post-test 9 month follow-up/post test & Interlock Ignition Device
  Interventions: Behavioral: Usual and Customary Information Group
- B-SMART Intervention Group (Experimental): Study Cohort Assessment:
  Baseline Web App Intervention 3 month follow-up/ post-test 9 month follow-up/post test & Interlock Ignition Device
  Interventions: Behavioral: B-SMART Intervention Group

INTERVENTIONS:
Behavioral: B-SMART Intervention Group — The B-SMART mobile web app will contain four modules: 1) Supporting Abstinence, 2) Shared Positive Activities, 3) Common Challenges for Family Members with IID, and 4) Effective Communication. Within each module there will be a series of learning activities, including presentation text, interactive engagement, and videos. All app content will be available in both English and Spanish, based on user language preference.
  Arms: B-SMART Intervention Group
Behavioral: Usual and Customary Information Group — Participants randomized to the usual and customary care (UC) group will receive a website with a pamphlet on the IID installed in their vehicle and the manufacturer information provided about the IID in PDF format, in both English and Spanish. This constitutes a UC group, as such pamphlets are widely available to DWI offenders who have IIDs installed in their vehicles. Thus, providing this pamphlet represents a standard information provision for first-time DWI offenders and their CFMs.
  Arms: Usual & Customary Information Group

SUMMARY:
The smart phone application (B-SMART) to be developed in this research project for family members of DWI (Driving While Intoxicated) offenders and offenders themselves will extend the impact of the Ignition Interlock Device (IID) and help DWI offenders and their families avoid drunk driving once the IID is removed from their automobiles. As such, the public health consequences of DWI, in terms of health, morbidity and mortality, and its economic and societal consequences, will be positively influenced by a highly accessible and diffusible intervention. The proposed Phase II project will complete the development and programming of the B-SMART smartphone web app and test its impact in a randomized efficacy trial with first-time DWI offenders and their concerned family members.

DETAILED DESCRIPTION:
Driving while intoxicated (DWI) remains a substantial and preventable source of morbidity and mortality in the United States. A variety of sanctions and interventions have been attempted to reduce DWI in the U.S., including enhanced DWI enforcement efforts, stricter drunk driving laws, responsible alcohol beverage service training, and alcohol treatment. The Ignition Interlock Device (IID), which requires a driver to blow into a breathalyzer unit installed in an automobile to establish sobriety, reduces drunk driving while installed. The use of IIDs has become widespread: most states in the U.S. now require convicted drunk drivers to install an IID in their cars upon some form of conviction. However, research has conclusively shown that once the IIDs are removed from DWI offenders' cars, DWI recidivism levels return to those comparable to offenders who did not have an IID. Interventions are needed to increase the likelihood that the effectiveness of IIDs persists beyond the installation period. The Brief Family-Involved Treatment (B-FIT) is a promising intervention to improve DWI recidivism by affecting the social environment of DWI offenders. Proposed here is Phase II research, a continuation of the original Phase I project, that will complete the translation of B-FIT into the B-SMART mobile web app for smartphones. The content of the intervention will be based on empirically-validated couples therapy for those with alcohol use disorders developed by Co-Investigator McCrady, translated to a smartphone platform. Phase II of this project will involve the systematic completion of B-SMART, employing: 1) an Expert Advisory Board, and 2) iterative development, multimedia and usability focus groups, and interviews comprised of CFM and DWI offenders. B-SMART will be fully produced for DWI offenders and their concerned family members (CFM) and then tested in a randomized controlled efficacy trial with first-time DWI offenders (n=150) and their CFMs (n=150) recruited from the Santa Fe County DWI Program. Unique to this intervention are the involvement of family members in supporting the DWI offender to not drink and drive and the use of smartphone technology to make that support immediate, accessible, and diffusible. B-SMART will involve the CFMs by providing coping skills, communication skills, and strategies to help avoid DWI. The randomized efficacy trial of B-SMART will examine B-SMART's impact on a variety of alcohol-related dependent variables, including IID lockout events, alcohol use, and family functioning. Should B-SMART be demonstrated to impact DWI offenders and their family members by reducing IID Lockout Events (which predict future DWI recidivism) and alcohol use, and improving family functioning, DWI offenders, their families, and their communities will have an important, effective, accessible tool to further reduce the social, health and economic consequences of DWI.

ELIGIBILITY:
Inclusion Criteria:

DWI Offender

* male or female
* 21 years or older
* first-time DWI offender with IID installed in vehicle
* enrolled in Santa Fe County DWI Program
* have a smartphone, tablet computer, or personal computer with Internet access
* consent to participate
* able to read and speak English or Spanish

Concerned Family Member (CFM):

* male or female
* 21 years or older
* spouse, parent, or immediate family member of first-time DWI offender with IID installed in vehicle and enrolled in Santa Fe County DWI Program
* have a smartphone, tablet computer, or personal computer with Internet access
* consent to participate
* able to read and speak English or Spanish

Exclusion Criteria:

* other family members already enrolled in the project
* second or above DWI conviction

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2019-03-30 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gill Woodall, PhD, Principal Investigator — Klein Buendel, Inc.
Locations (2):
- United States (2):
  - Klein Buendel, Inc, Golden, Colorado
  - University of New Mexico, Albuquerque, New Mexico

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual & Customary Information Group: Study Cohort Assessment:
  Baseline 3 month follow-up/ post-test 9 month follow-up/post test & Interlock Ignition Device
  Usual and Customary Information Group: Participants randomized to the usual and customary care (UC) group will receive a website with a pamphlet on the IID installed in their vehicle and the manufacturer information provided about the IID in PDF format, in both English and Spanish. This constitutes a UC group, as such pamphlets are widely available to DWI offenders who have IIDs installed in their vehicles. Thus, providing this pamphlet represents a standard information provision for first-time DWI offenders and their CFMs.
- B-SMART Intervention Group: Study Cohort Assessment:
  Baseline Web App Intervention 3 month follow-up/ post-test 9 month follow-up/post test & Interlock Ignition Device
  B-SMART Intervention Group: The B-SMART mobile web app will contain four modules: 1) Supporting Abstinence, 2) Shared Positive Activities, 3) Common Challenges for Family Members with IID, and 4) Effective Communication. Within each module there will be a series of learning activities, including presentation text, interactive engagement, and videos. All app content will be available in both English and Spanish, based on user language preference.
Period: Baseline
Arm/Group | Usual & Customary Information Group | B-SMART Intervention Group
Started | 130 | 116
Completed | 130 | 116
Not Completed | 0 | 0
Period: 3 Month Follow-up
Arm/Group | Usual & Customary Information Group | B-SMART Intervention Group
Started | 130 | 116
Completed | 126 | 104
Not Completed | 4 | 12
Not completed — Lost to Follow-up | 4 | 12
Period: 9 Month Follow up
Arm/Group | Usual & Customary Information Group | B-SMART Intervention Group
Started | 126 | 104
Completed | 114 | 84
Not Completed | 12 | 20
Not completed — Lost to Follow-up | 12 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual & Customary Information Group | B-SMART Intervention Group | Total
Number analyzed (Participants) | 130 | 116 | 246
Age, Continuous [Mean (Standard Deviation); unit: years] — Years of Age of Participants
  years | 38.96 (13.39) | 38.09 (13.42) | 38.55 (13.38)
Sex: Female, Male [Count of Participants; unit: Participants] — Self Report of Gender at Birth
  Participants
    Female | 77 | 62 | 139
    Male | 53 | 54 | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 70 | 50 | 120
  Not Hispanic or Latino | 49 | 48 | 97
  Unknown or Not Reported | 11 | 18 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 15 | 19 | 34
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
  Black or African American | 4 | 4 | 8
  White | 67 | 54 | 121
  More than one race | 6 | 2 | 8
  Unknown or Not Reported | 35 | 37 | 72

OUTCOME MEASURES:

1. Primary Outcome: Measure of Primary Outcome Variable: IID Lockout Events.
Description: The primary outcome measure will be frequency of IID lockout events from baseline to 9-month follow-up post-randomization, collected from Ignition Interlock providers for participants in the study design. Lockout events occur on an Ignition Interlock Device when a user repeatedly fails a breathalyzer test within a given time frame to allow the automobile to start. When a user repeatedly fails the IID test, the device locks out the automobile's ignition, thus a Lockout Event occurs. These events are significant in that they indicate an attempt by the user to drive while intoxicated. In prior research Lockout Events predict subsequent DWI recidvism.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: Ignition Interlock Lockout Events
Arm/Group | Usual & Customary Information Group | B-SMART Intervention Group
Number analyzed (Participants) | 45 | 26
Ignition Interlock Lockout Events | 10.13 (18.34) | 2.78 (5.06)
Statistical Analysis 1: Comparison: Usual & Customary Information Group vs B-SMART Intervention Group; Test type: Superiority; p = .04, ANOVA

2. Secondary Outcome: Measures of Secondary Outcome Variables and Mediators.
Description: Alcohol use by the DWI offender, a secondary outcome, will be assessed at baseline, 3-month follow-up, and 9-month follow-up with versions of the Form 9090,91 adapted for online assessment for the CFMs (Form 90-ACS) and first-time DWI offenders (Form 90-AF).
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual & Customary Information Group | B-SMART Intervention Group
Number analyzed (Participants) | 57 | 42
Participants | 20 | 7
Statistical Analysis 1: Comparison: Usual & Customary Information Group vs B-SMART Intervention Group; Test type: Superiority; p = .034, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected over a 9-month period for each participant.
Arm/Group | Usual & Customary Information Group | B-SMART Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/130 | 0/116
Serious Adverse Events (participants affected / at risk) | 0/130 | 0/116
Other Adverse Events (participants affected / at risk) | 0/130 | 0/116

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT03828370/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT03828370/ICF_001.pdf